CLINICAL TRIAL: NCT04941469
Title: Effectiveness of Specifically Optimized Off-the-counter Foot Orthosis for the Management of Mechanical Foot Pains in the Subtle Cavus Foot Type: A Pilot-controlled Study
Brief Title: Effectiveness of Specifically Optimized Off-the-counter Foot Orthosis for the Subtle Cavus Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Ng Chuan Guan, Senior Podiatrist, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/01043
Record Dates: First submitted 2021-06-14; First posted 2021-06-28 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Subtle Cavus Foot; Mechanical Foot Pains; Plantar Fasciitis; Achilles Tendinopathy; Insertional Achilles Tendinopathy; Strain of Peroneal Tendon; Metatarsalgia; Pes Cavus; Pes Cavus, Bilateral; Pes Cavovarus
Keywords: Mechanical foot pains; Prefabricated insoles; Off the counter insoles; Optimized insoles
MeSH Terms: conditions — Fasciitis, Plantar; Metatarsalgia; Talipes Cavus

STUDY DESIGN:
Intervention Model Description: This is a Pilot Randomized Controlled Trial designed to compare the effectiveness of specifically optimized off-the-counter foot orthosis versus plain off-the-counter foot orthosis in managing mechanical foot pains in the Subtle Cavus foot type
  * Subjects recruited will be randomly assigned to either the plain off-the-counter foot orthosis group (Control Group) or the specifically optimized off-the-counter foot orthosis group (Intervention Group) based on a pre-specified randomization list during the Screening Visit.
  * Randomization was performed using the Randomized Permuted Block Randomization method with blocks of six.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specifically optimized off-the-counter foot orthosis (Experimental): The study device is a specifically optimized off-the-counter foot orthosis modified by an additional wedging added onto the original Formthotics (Original Dual Hard) with standard arch fill reduction to achieve a foot orthosis that is "tailored" for the management of mechanical foot pains in the Subtle Cavus foot type.
  Interventions: Device: Specifically optimized off-the-counter foot orthosis (Medical grade foot orthosis)
- Plain off-the-counter foot orthosis (Active Comparator): The control device for this study would be the plain original Formthotics (Original Dual Hard).
  Interventions: Device: Plain off-the-counter foot orthosis (Medical grade foot orthosis)

INTERVENTIONS:
Device: Specifically optimized off-the-counter foot orthosis (Medical grade foot orthosis) — The study device is a specifically optimized off-the-counter foot orthosis modified by an additional wedging added onto the original Formthotics (Original Dual Hard) with standard arch fill reduction to achieve a foot orthosis that is "tailored" for the management of mechanical foot pains in the Subtle Cavus foot type. The original Formthotics (Original Dual Hard) is currently in use and is considered a Class A medical device according to the Health Science Authority of Singapore risk classification system. At the moment, the original Formthotics (Original Dual Hard) is also available in the retail market, abeit, without assessment guided optimisations for specific feet types.
  Other Names: Specifically optimized prefabricated foot orthosis; Specifically optimized prefabricated Insoles
  Arms: Specifically optimized off-the-counter foot orthosis
Device: Plain off-the-counter foot orthosis (Medical grade foot orthosis) — The control device for this study would be the plain original Formthotics (Original Dual Hard).
  Other Names: Plain prefabricated foot orthosis; Plain prefabricated Insoles
  Arms: Plain off-the-counter foot orthosis

SUMMARY:
As off-the-counter foot orthoses are readily available and have an economic advantage, they are increasingly being used by healthcare professionals to treat mechanical foot pains in place of custom foot orthosis. However, there is a lack of available evidence to determine if a plain off-the-counter foot orthosis that aims to contours to the foot or a specifically optimized off-the-counter foot orthosis utilizing the type of orthotic design proposed by Abbasian and Pomeroy is more effective in the management of mechanical foot pains in the Subtle Cavus foot type.

This study proposal seeks to fill the gap in this area.

Primary Aim:

To investigate the effectiveness of specifically optimized off-the-counter foot orthosis designed for the Subtle Cavus foot type in improving patient reported outcomes in patients with mechanical foot pains when compared to plain off-the-counter foot orthosis.

Primary Null Hypothesis:

There is no difference in pain and functional scores reported by patients between specifically optimized off-the-counter foot orthosis and plain off-the-counter foot orthosis in patients with mechanical foot pains at four, eight and twelve weeks of intervention.

In our study, the Subtle Cavus foot refers to the flexible idiopathic forefoot-driven Pes Cavus that can be clinically recognised with a positive "Peek a Boo" sign, inverted hindfoot position in weight bearing stance and Positive Coleman Block Test as reported by Manoli and Graham in 2005.

Also, for our study, mechanical foot pains are limited to clinically diagnosed Plantar Fasciitis, Achilles Tendinopathy, Peroneal Strain or Metatarsalgia:

Plantar Fasciitis is clinically diagnosed using the following history and physical examination findings:

* Plantar medial heel pain /or pain along the plantar fascia: most noticeable with initial steps after a period of inactivity but also worse following prolonged weight bearing
* Heel pain /or pain along the plantar fascia precipitated by a recent increase in weightbearing activity
* Pain with palpation of the proximal insertion of the plantar fascia /or along the band of plantar fascia structure

Achilles Tendinopathy is clinically diagnosed using the following history and physical examination findings:

Midportion Achilles Tendinopathy:

* Self-reported localized pain and perceived stiffness in the Achilles tendon following a period of inactivity (eg, sleep, prolonged sitting) lessen with an acute bout of activity and may increase after the activity.
* Symptoms are frequently accompanied by Achilles tendon tenderness.
* Pain located 2 to 6 cm proximal to the Achilles tendon insertion that began gradually and pain with palpation of the midportion of the tendon to diagnose midportion Achilles tendinopathy

Insertional Achilles Tendinopathy:

* Self-reported pain that is aggravated by activity and stiffness that is associated with prolonged periods of rest.
* Pain and tenderness with palpation within the distal 2 cm of the Achilles tendon.
* Redness and swelling over area of Achilles Tendon insertion over posterior heel

Peroneal Strain is clinically diagnosed using the following history and physical examination findings:

* Pain and swelling posterior to the lateral malleolus
* Pain with active eversion and dorsiflexion against resistance
* May have a history of chronic lateral ankle pain and instability
* Pain and tenderness with palpation along the course of the peroneal tendons

Metatarsalgia is clinically diagnosed using the following history and physical examination findings:

* Self-reported pain during the propulsive phase of gait. The pain is localized underneath the prominent metatarsal heads
* The plantar soft tissue can be swollen and inflamed.
* Presence of hyperkeratosis over tender areas may be present
* Pain and tenderness with palpation of plantar metatarsophalangeal joints

Secondary Aim:

To investigate the effectiveness of specifically optimized off-the-counter foot orthosis designed for the Subtle Cavus foot type in improving patient reported outcomes in patients with mechanical foot pains pre- and post-intervention.

Secondary Null Hypothesis:

There is no difference in pain and functional scores reported by patients after introduction of specifically optimized off-the counter foot orthosis pre- and post-intervention at initial to four, initial to eight and initial to twelve weeks of intervention.

DETAILED DESCRIPTION:
Study Design:

This is a Pilot Randomized Controlled Trial designed to compare the effectiveness of specifically optimized off-the-counter foot orthosis versus plain off-the-counter foot orthosis in managing mechanical foot pains in the Subtle Cavus foot type. (See Figure 3).

* Subjects recruited will be randomly assigned to either the plain off-the-counter foot orthosis group (Control Group) or the specifically optimized off-the-counter foot orthosis group (Intervention Group) based on a pre-specified randomization list during the Screening Visit.
* Randomization was performed using the Randomized Permuted Block Randomization method with blocks of six.
* For participants with bilateral mechanical foot pains, the more symptomatic side will be used as the reference for collection of participants reported outcome measures throughout the study.
* There will be an intervention period of 12 weeks, which is a common therapy window for the associated symptoms of mechanical foot pains.
* All other standard of care Podiatry management will be implemented for all subjects in the two groups throughout the study period.
* Standard Podiatry management with stretching exercise regime refers to the following protocols with official department stretching and strengthening brochure provided for all subjects:

Towel Stretch (To be introduced at Study Visit 1 (Week 0)):

Sit down and extend both legs Pass a towel around the top of your foot Slowly pull the towel towards your body Hold each stretch for a period of 20 seconds Switch sides and repeat Repeat the stretch 10 times on both sides for each set Perform 2 sets a day

Gastrocnemius Stretch (To be introduced at Study Visit 2 (Week 4)):

Place both hands on a wall and stand an arm's length away from it Place one foot behind the other Bend your front knee Ensure your back knee and back are straight Ensure both heels are flat on the floor Do not rotate your hips Ensure both feet are parallel Hold each stretch for a period of 20 seconds Switch legs and repeat Repeat the stretch 10 times on both sides for each set Perform 2 sets a day

Soleus Stretch (To be introduced at Study Visit 2 (Week 4)):

Place both hands on a wall and stand an arm's length away from it Place one foot behind the other Bend both knees Keep both heels flat on the floor Ensure your back is straight Do not rotate your hips Ensure both feet are parallel Hold each stretch for a period of 20 seconds Switch legs and repeat Repeat the stretch 10 times on both sides for each set Perform 2 sets a day

Double Leg Tip Toe (To be introduced at Study Visit 3 (Week 8)):

With both knees straight, go up on tiptoes on both feet (A) Gently lower both heels to the ground (B) Repeat 10 times Perform 2 sets a day

* Standard Podiatry management for foot orthosis troubleshooting refers to: Bilateral Standard Arch Fill Reduction of foot orthoses if study participant complains of discomfort / irritation from use of foot orthosis over the arches of the feet for both plain off-the-counter foot orthosis or specifically optimised off-the-counter foot orthosis.
* Subjects' pain and functional impairment perception will be measured pre- and post-intervention at Study Visit 1 (Week 0), Study Visit 2 (Week 4), Study Visit 3 (Week 8) and the Study Visit 4 (Week 12).
* Participants will also be asked regarding compliance towards the use of the foot orthosis fitted and other standard podiatry management that has been started and Patient Satisfaction Ratings with Podiatry Treatment introduced using a verbal compliance ratings form administered by the investigators during Study Visit 2 (Week 4), Study Visit 3 (Week 8) and Study Visit 4 (Week 12).
* Outcome measures of the specifically optimized off-the-counter foot orthosis group will be compared against the plain off-the-counter foot orthosis group to achieve the primary aim of the study.
* Pre and post intervention within group comparison of outcome measures will be conducted for both groups independently to achieve the secondary aim of the study.

Outcome measures:

Primary outcome measure:

* The Foot Function Index (FFI) total score
* The FFI is a self-reported measure of pain, function, and activity level associated with foot dysfunction consisting of 23 items divided into 3 sub-scales. The scores range from 0 to 10, with the higher scores indicating more disability.
* The FFI has been validated and is recommended as a reliable measurement scale for use in foot orthotic interventions study.
* The evaluation of the study device efficacy will be conducted with the main outcome measure, the FFI, before and after the intervention.

Secondary outcome measure:

* The FFI sub-scale scores in the domain of pain, disability and activity limitation
* The subscales of the FFI will be analysed separately as secondary outcome measures.

Tertiary outcome measure:

* 100mm Visual Analogue Scale (VAS) with the end-points "no pain" and "worst pain possible"
* It is a reliable and valid measure of self-reported pain intensity
* VAS is administered before and after intervention to evaluate acute pain levels

Study Setting:

Podiatry outpatient clinic at Foot Care and Limb Design Centre, Tan Tock Seng Hospital.

Study Population:

Study population will be drawn from the patients referred to Podiatry Department, Foot Care and Limb Design Centre, Tan Tock Seng Hospital for Biomechanics Assessment.

* Adult patients with clinically diagnosed mechanical foot pains limited to Plantar Fasciitis, Achilles Tendinopathy, Peroneal Strain or Metatarsalgia will be eligible.
* For participants with bilateral mechanical foot pains, the more symptomatic side will be used as the reference for collection of participants reported outcome measures throughout the study.
* There is no subject restriction based on the race of the subjects.

Standard Podiatry clinical assessments and a full biomechanical assessment will be performed to determine eligibility of potential study participants.

1. Clinical diagnoses of mechanical foot pains limited to Plantar Fasciitis, Achilles Tendinopathy, Peroneal Strain or Metatarsalgia will be done through Physical / Clinical assessments.
2. For participants with bilateral mechanical foot pains, the more symptomatic side will be used as the reference for collection of participants reported outcome measures throughout the study.
3. Subtle cavus foot type will be identified through a full biomechanical assessment including the "Peek a boo" sign and the Coleman Block Test.
4. Inclusion and Exclusion criteria will be checked against when the above two conditions are met.

On top of outcome measure questionnaires that will be administered, Study team will retrieve data from participant's medical records including basic demographics, standard podiatry assessments results and management measures and outcomes as well. These data will be recorded into the study database document provided.

There will not be any incidental findings arising in this research.

Sample size calculation for comparison between two independent means and paired means:

Taking a 7-point difference in FFI total score as clinically significant / minimal important difference:

* Alpha error = 0.05
* Power (1-beta error) = 0.80
* Two-tailed Test
* Difference in mean = 7
* Standard Deviation in each group = 7

Required Sample size is estimated to be at least 16 or more in each group. Hence, target at least 20 in each group taking into consideration drop-out and lost to follow-up.

Taking a 12-point difference in FFI pain sub-scale score as clinically significant / minimal important difference:

* Alpha error = 0.05
* Power (1-beta error) = 0.80
* Two-tailed Test
* Difference in mean = 12
* Standard Deviation in each group = 12

Required Sample size is estimated to be at least 16 or more in each group. Hence, target at least 20 in each group taking into consideration drop-out and lost to follow-up.

Taking a 7-point difference in FFI disability sub-scale score as clinically significant / minimal important difference:

* Alpha error = 0.05
* Power (1-beta error) = 0.80
* Two-tailed Test
* Difference in mean = 7
* Standard Deviation in each group = 7

Required Sample size is estimated to be at least 16 or more in each group. Hence, target at least 20 in each group taking into consideration drop-out and lost to follow-up.

Taking a 9mm difference in 100mm VAS pain score as clinically significant / minimal important difference:

* Alpha error = 0.05
* Power (1-beta error) = 0.80
* Two-tailed Test
* Difference in mean = 9
* Standard Deviation in each group = 9

Required Sample size is estimated to be at least 16 or more in each group. Hence, target at least 20 in each group taking into consideration drop-out and lost to follow-up.

Reference:

1. R Core Team (2020). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL https://www.R-project.org/
2. Landorf KB, Radford JA (2008): Minimal important difference: values for the foot health status questionnaire, foot function index and visual analogue scale. The Foot, 18(1): 15-19.

Statistical and Analytical Plans:

Baseline data such as Age, Gender, Ethnicity, pre-intervention outcome measures and other data collected will be explored to determine data distribution and whether data fit a normal distribution using the Shapiro-Wilk Test. Other exploration such as Q-Q plot visual inspection will be utilised also.

The Independent Student t-test for comparison between two means for FFI total score, FFI pain sub-scale score, FFI disability sub-scale score and VAS pain score between specifically optimized off-the-counter foot orthosis and plain off-the-counter foot orthosis at zero, four, eight and twelve-weeks post intervention will be utilised.

Pre- and post-intervention within group comparison will also be analysed using the Paired t-test for both the specifically optimized off-the-counter foot orthosis group and the plain off-the-counter foot orthosis group at initial to four, initial to eight and initial to twelve weeks of intervention.

Minimal important difference for all outcome measures such as the FFI total score, FFI pain sub-scale score, FFI disability sub-scale score and VAS pain score are based on the values reported by Landorf and Radford in 2008.

Statistical significance is defined at the 5% (P = 0.05) level as determined above.

Non-parametric statistical methods such as the Wilcoxon signed rank test and Wilcoxon rank sum test may be applied accordingly if exploratory analysis show that the distribution of data collected is skewed.

Data analysis software that will be applied:

* R from R Foundation for Statistical Computing, Vienna, Austria
* R Core Team (2020). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL https://www.R-project.org/

Procedures/ activities that are carried out for the purpose of research:

Screening Visit:

Potential participants will be assessed by the Principal Investigator or the Co-Investigator to identify if they are eligible to participate in the study. If the subject fit the inclusion criteria, the on-site investigator will provide an information package, and explain and obtain written consent. Subject will be encouraged to ask any questions regarding the study.

If the participant consent to take part in the study, his/her demographics, medical and clinical data will be obtained from their medical records at Foot Care and Limb Design Centre at Tan Tock Seng Hospital. Participants will be randomly assigned to receive either specifically optimized off-the-counter foot orthosis or plain off-the-counter foot orthosis based on a pre-specified randomization list upon enrolment into the study. Clinical foot orthosis measurement for either a pair of plain off-the-counter foot orthosis or a pair of specifically optimized off-the-counter foot orthosis suitable for subject's feet will be provided.

Study Visit 1 (Week 0) Research participants will be fitted with either the specifically optimized off-the-counter foot orthosis or plain off-the-counter foot orthosis on Study Visit 1 (Week 0) as assigned during the Screening Visit.

Study Visit 1 to 4 (Week 0 to Week 12) Collection of patient reported outcome measures such as The Foot Function Index (FFI) total score and its sub-scale scores in the domain of pain, disability and activity limitation and the 100mm Visual Analogue Scale (VAS) with the end-points "no pain" and "worst pain possible" for the purpose of research will be carried out.

All patient reported outcome measures will be collected at Study visit 1(week 0), Study Visit 2 (week 4), Study visit 3 (Week 8) and Study Visit 4 (week 12).

Study Visit 2 to 4 (Week4 to Week 12) Collection of patient reported Verbal Compliance Ratings towards the use of the foot orthosis fitted and other standard podiatry management using a verbal compliance ratings form administered by the investigators during the study visit will be carried out.

All patient reported Verbal Compliance Ratings will be collected at Study Visit 2 (week 4), Study visit 3 (Week 8) and Study Visit 4 (week 12).

Study Visit 2 to 4 (Week4 to Week 12) Collection of Patient Satisfaction Ratings using a verbal compliance ratings form administered by the investigators during the study visit will be carried out.

All Patient Satisfaction Ratings will be collected at Study Visit 2 (week 4), Study visit 3 (Week 8) and Study Visit 4 (week 12).

Activities that are performed for routine diagnostic or standard medical treatment as part of the research participant's standard care:

Screening visit Standard Podiatry Biomechanical assessment to determine the participant's biomechanics profile is performed as part of standard care. Standard appropriate footwear advice (neutral running sport shoes as labelled by the retail manufacturers such as New Balance 880, Asics Nimbus, etc.) for the fitting of subject's foot orthosis at the next follow-up visit will be provided as part of standard care. Participants will receive standard best practice Podiatry treatment for their mechanical foot pains.

Study Visit 1 (Week 0) The subject will be required to return to Foot Care and Limb Design Centre for follow-up consultation with a pair of neutral running sport shoes for fitting of either a specifically optimized off-the-counter foot orthosis or plain off-the-counter foot orthosis that has been pre-assigned during the screening visit. Standard Podiatry assessment and routine management will be provided which includes introduction of clinically indicated stretching exercise regime and foot orthosis troubleshooting. Participant will receive standard best practice Podiatry treatment for their mechanical foot pains.

Study Visit 2 (Week 4) The subject will be required to return to Foot Care and Limb Design Centre for follow-up consultation with a pair of neutral running sport shoes and foot orthosis that has been fitted previously. Standard Podiatry assessment and routine management will be provided which includes introduction and review of clinically indicated stretching exercise regime and foot orthosis troubleshooting. Participant will receive standard best practice Podiatry treatment for their mechanical foot pains.

Study Visit 3 (Week 8) The subject will be required to return to Foot Care and Limb Design Centre for follow-up consultation with a pair of neutral running sport shoes and foot orthosis that has been fitted previously. Standard Podiatry assessment and routine management will be provided which includes introduction and review of clinically indicated stretching exercise regime and foot orthosis troubleshooting. Participant will receive standard best practice Podiatry treatment for their mechanical foot pains.

Study Visit 4 (Week 12) The subject will be required to return to Foot Care and Limb Design Centre for follow-up consultation with a pair of neutral running sport shoes and foot orthosis that has been fitted previously. Standard Podiatry assessment and routine management will be provided which includes introduction and review of clinically indicated stretching exercise regime and foot orthosis troubleshooting. Participant will receive standard best practice Podiatry treatment for their mechanical foot pains

Potential Benefits (direct as well as indirect) to research participants and to the society:

Direct Benefits:

Study participant may reasonably expect to benefit from the trial's specifically optimized off-the-counter foot orthosis or plain off-the-counter foot orthosis in the following way: The study device providing optimal biomechanical control leading to reduce stress over injured structures of the feet which typically translate to symptoms or pain reduction for the user.

Indirect shorter-term Benefits:

This study will provide evidence for or against the use of specifically optimized off-the-counter foot orthosis in the management of mechanical foot pains in the Subtle Cavus foot type. The findings of this study will help to build up knowledge in foot orthotic therapy delivery. If specifically optimized off-the-counter foot orthosis is proven more effective than plain off-the-counter foot orthosis, this can provide evidence to support the use of assessment directed foot orthosis prescription as in the case of utilising the Coleman Block Test to differentiate between flexible forefoot-driven Subtle Cavus foot type from a hindfoot driven Rigid Pes Cavus foot type compared to a "generic" foot orthosis that simply contours to the arch of the foot.

As the optimisations suggested are specific, this will help practitioners to confidently apply wedging techniques and perform standard arch fill reduction that can be consistently replicated. Furthermore, incidences of foot orthosis that are optimized wrongly will be reduced with standardized optimizations leading to better standard of care.

Specifically optimized off-the-counter foot orthosis which is "tailored" to the presenting Subtle Cavus foot type is cheaper than current custom solutions. If found to be effective when compared to a generic plain off-the counter foot orthosis, further research can be conducted to determine if a specifically optimized off-the-counter foot orthosis is as effective and non-inferior to a custom foot orthosis with the same specifications. As optimized off-the-counter foot orthosis can be readily fitted, foot orthotic therapy can be instituted without any delay. Improvement in treatment outcomes can be expected as patients will receive timely foot orthotic intervention.

If specifically optimized off-the-counter foot orthosis is as effective and non-inferior to a custom foot orthosis with the same specifications. It can provide an easily available, cost-effective foot orthosis for patients as custom foot orthosis are at least three times the cost of a specifically optimized off-the-counter foot orthosis and require at least two weeks for such a custom solution to be made.

In summary, this project has the potential to make podiatry care delivery for patients with painful Subtle Cavus foot type better, safer, faster and cheaper.

Indirect longer-term benefit:

Currently, foot orthosis construction for diabetic foot offloading in ulcer prevention is also based on the principle of increasing contact area to reduce pressure at a particular point. The findings of this study can potentially help to understand how offloading of the diabetic foot in ulcer prevention can be relooked for the Subtle Cavus foot type. If specifically optimized off-the-counter foot orthosis is proven to be more effective than plain off-the-counter foot orthosis in managing mechanical foot pains in the Subtle Cavus foot type, this can provide evidence to further investigate if specifically optimised off-the-counter foot orthosis can perform better than a device that simply contours to the foot in diabetic offloading for ulcer prevention. A cheaper and faster "tailored" solution like specifically optimised off-the-counter foot orthosis can benefit patient care in the long run in offloading the diabetic foot.

With emerging technology such as data analytics and machine learning, this project may potentially lay the foundation to spur further research in the area of feet type recognition for the Subtle Cavus foot type and the Pes Planus foot type using visual analytics techniques.

Safety Monitoring plan, i.e. frequency of review (e.g. daily, weekly, quarterly) and type of data (e.g. adverse events/serious adverse events) will be monitored:

Frequency of review: Monthly at every study visit on Study visit 1, Study visit 2, Study visit 3 and the Final Visit.

Adverse events or Serious adverse events will be monitored

Assessment plan:

A standard physical examination of the feet will be conducted at every study visit on Study visit 1, Study visit 2, Study visit 3 and the Final Visit.

Description of anticipated events including character and expected incidence:

1. Study participant complaining of discomfort / irritation from use of foot orthosis over plantar aspect of the feet (both conventional custom foot orthosis or specifically optimised off-the-counter foot orthosis) Such incidences can happen and are expected in routine and standard foot orthotic therapy in about 30% of users based on PI's clinical experience. It is also expected that some people might need longer period of time to get used to foot orthotic therapy. Simple trouble shooting of foot orthosis can resolve the complaint most of the time.
2. Study participant complaining of intolerance to foot orthosis use and are not able to continue wearing the device even after simple trouble shooting of foot orthosis has been provided.

Such incidence can happen and are expected in routine and standard foot orthotic therapy in about less than 5% of users based on PI's clinical experience. Study participant will be advised to stop foot orthotic therapy.

3/4. Rarely, the use of foot orthosis can cause more mechanical pains or create friction between the device and the sole of the feet resulting in blister formation. Symptoms of such occurrences include: increased pain when using the device but has no issues when not using the device, redness over the arch area or blister formation. If participants have any of these symptoms, they will be advised to stop the use of the device immediately and to call the Podiatrist or principal investigator at once.

Plan for grading the seriousness of events:

1. Discomfort / Irritation from foot orthosis use
2. Intolerance to foot orthosis use
3. Friction between foot orthosis and plantar sole of foot resulting in rubbing and redness
4. Friction between foot orthosis and plantar sole of foot resulting in blister formation

Both 1 and 2 can be considered expected incidences in standard foot orthotic therapy and does not amount to an adverse event.

Both 3 and 4 can be considered adverse events not amounting to serious adverse events.

Plan for assessing the causal relationship of events to the study:

For both 1 and 2, standard simple troubleshooting of foot orthosis will be rendered to assess for causal relationship. If discomfort / irritation / intolerance is resolved, there is a possible causal relationship between events 1 and 2 to the study device being investigated.

For 3 and 4, study participant will be advised to stop the use of the study device until redness or blister has resolved prior to restarting foot orthotic therapy again (with simple trouble shooting of foot orthosis rendered). If redness or blister formation is resolved, there is a possible causal relationship between events 3 or 4 to the study device being investigated.

Data monitoring will be done in accordance with ICH GCP by the PI on a quarterly basis to ensure data integrity is assured.

Route of dissemination of any data and safety information to the study sites, as well as the person/team responsible for doing so:

PI will conduct monthly face-to-face ad-hoc meetings to discuss and update data and safety information with the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21-80 years old
2. Able to provide informed consent
3. Clinically diagnosed mechanical foot pains limited to Plantar Fasciitis, Achilles Tendinopathy, Peroneal Strain or Metatarsalgia.
4. Clinically recognized Subtle Cavus foot type
5. Positive "Peek a boo" sign
6. Hind foot / Rearfoot / Heel in varus position in weight bearing stance
7. Positive Coleman Block Test (rearfoot inversion correctable)
8. Able to comply with all study procedures

Exclusion Criteria:

1. Age < 21 Years old
2. History of surgery in the lower limb
3. History of trauma or falls prior to onset of symptoms or after
4. Pregnancy or breastfeeding women
5. Pes Planus foot type
6. Rigid Pes Cavus (Negative Coleman Block Test)
7. Nervous system problems (e.g., stroke, dementia, seizures)
8. Peripheral vascular pathology
9. Acute infection
10. Rheumatic joint disease
11. Inability to comply to wearing appropriate footwear and foot orthosis
12. Lack of willingness to return for follow-up
13. Musculoskeletal pathology other than Plantar Fasciitis, Achilles Tendinopathy, Peroneal Strain or Metatarsalgia

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
The Foot Function Index (FFI) total score | Study Visit 2 (Week 4)
  * The FFI is a self-reported measure of pain, function, and activity level associated with foot dysfunction consisting of 23 items divided into 3 sub-scales. The scores range from 0 to 10, with the higher scores indicating more disability.
  * The FFI has been validated and is recommended as a reliable measurement scale for use in foot orthotic interventions study.
  * The evaluation of the study device efficacy will be conducted with the main outcome measure, the FFI between the control and treatment groups.
The Foot Function Index (FFI) total score | Study Visit 3 (Week 8)
  * The FFI is a self-reported measure of pain, function, and activity level associated with foot dysfunction consisting of 23 items divided into 3 sub-scales. The scores range from 0 to 10, with the higher scores indicating more disability.
  * The FFI has been validated and is recommended as a reliable measurement scale for use in foot orthotic interventions study.
  * The evaluation of the study device efficacy will be conducted with the main outcome measure, the FFI between the control and treatment groups.
The Foot Function Index (FFI) total score | Study Visit 4 (Week 12)
  * The FFI is a self-reported measure of pain, function, and activity level associated with foot dysfunction consisting of 23 items divided into 3 sub-scales. The scores range from 0 to 10, with the higher scores indicating more disability.
  * The FFI has been validated and is recommended as a reliable measurement scale for use in foot orthotic interventions study.
  * The evaluation of the study device efficacy will be conducted with the main outcome measure, the FFI between the control and treatment groups.
The Change in Foot Function Index (FFI) total score from baseline at Week 4 | Study Visit 2 (Week 4) vs Study Visit 1 (Week 0)
  * The FFI is a self-reported measure of pain, function, and activity level associated with foot dysfunction consisting of 23 items divided into 3 sub-scales. The scores range from 0 to 10, with the higher scores indicating more disability.
  * The FFI has been validated and is recommended as a reliable measurement scale for use in foot orthotic interventions study.
  * The evaluation of the study device efficacy will be conducted with the main outcome measure, the FFI before and after intervention.
The Change in Foot Function Index (FFI) total score from baseline at Week 8 | Study Visit 3 (Week 8) vs Study Visit 1 (Week 0)
  * The FFI is a self-reported measure of pain, function, and activity level associated with foot dysfunction consisting of 23 items divided into 3 sub-scales. The scores range from 0 to 10, with the higher scores indicating more disability.
  * The FFI has been validated and is recommended as a reliable measurement scale for use in foot orthotic interventions study.
  * The evaluation of the study device efficacy will be conducted with the main outcome measure, the FFI before and after intervention.
The Change in Foot Function Index (FFI) total score from baseline at Week 12 | Study Visit 4 (Week 12) vs Study Visit 1 (Week 0)
  * The FFI is a self-reported measure of pain, function, and activity level associated with foot dysfunction consisting of 23 items divided into 3 sub-scales. The scores range from 0 to 10, with the higher scores indicating more disability.
  * The FFI has been validated and is recommended as a reliable measurement scale for use in foot orthotic interventions study.
  * The evaluation of the study device efficacy will be conducted with the main outcome measure, the FFI before and after intervention.

SECONDARY OUTCOMES:
The FFI sub-scale scores in the domain of pain | Study Visit 2 (Week 4)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of pain between the control and treatment groups.
The FFI sub-scale scores in the domain of pain | Study Visit 3 (Week 8)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of pain between the control and treatment groups.
The FFI sub-scale scores in the domain of pain | Study Visit 4 (Week 12)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of pain between the control and treatment groups.
The FFI sub-scale scores in the domain of disability | Study Visit 2 (Week 4)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of disability between the control and treatment groups.
The FFI sub-scale scores in the domain of disability | Study Visit 3 (Week 8)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of disability between the control and treatment groups.
The FFI sub-scale scores in the domain of disability | Study Visit 4 (Week 12)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of disability between the control and treatment groups.
The FFI sub-scale scores in the domain of activity limitation | Study Visit 2 (Week 4)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of activity limitation between the control and treatment groups.
The FFI sub-scale scores in the domain of activity limitation | Study Visit 3 (Week 8)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of activity limitation between the control and treatment groups.
The FFI sub-scale scores in the domain of activity limitation | Study Visit 4 (Week 12)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of activity limitation between the control and treatment groups.
The Change in FFI sub-scale scores in the domain of pain from baseline at Week 4 | Study Visit 2 (Week 4) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of pain before and after intervention.
The Change in FFI sub-scale scores in the domain of pain from baseline at Week 8 | Study Visit 3 (Week 8) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of pain before and after intervention.
The Change in FFI sub-scale scores in the domain of pain from baseline at Week 12 | Study Visit 4 (Week 12) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of pain before and after intervention.
The Change in FFI sub-scale scores in the domain of disability from baseline at Week 4 | Study Visit 2 (Week 4) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of disability before and after intervention.
The Change in FFI sub-scale scores in the domain of disability from baseline at Week 8 | Study Visit 3 (Week 8) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of disability before and after intervention.
The Change in FFI sub-scale scores in the domain of disability from baseline at Week 12 | Study Visit 4 (Week 12) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of disability before and after intervention.
The Change in FFI sub-scale scores in the domain of activity limitation from baseline at Week 4 | Study Visit 2 (Week 4) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of activity limitation before and after intervention.
The Change in FFI sub-scale scores in the domain of activity limitation from baseline at Week 8 | Study Visit 3 (Week 8) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of activity limitation before and after intervention.
The Change in FFI sub-scale scores in the domain of activity limitation from baseline at Week 8 | Study Visit 4 (Week 12) vs Study Visit 1 (Week 0)
  - The evaluation of the study device efficacy will be conducted with the FFI sub-scale scores in the domain of activity limitation before and after intervention.
100mm Visual Analogue Scale (VAS) with the end-points "no pain" and "worst pain possible" | Study Visit 1 (Week 0)
  * It is a reliable and valid measure of self-reported pain intensity
  * VAS is administered before and after intervention to evaluate acute pain levels
100mm Visual Analogue Scale (VAS) with the end-points "no pain" and "worst pain possible" | Study Visit 2 (Week 4)
  * It is a reliable and valid measure of self-reported pain intensity
  * VAS is administered before and after intervention to evaluate acute pain levels
100mm Visual Analogue Scale (VAS) with the end-points "no pain" and "worst pain possible" | Study Visit 3 (Week 8)
  * It is a reliable and valid measure of self-reported pain intensity
  * VAS is administered before and after intervention to evaluate acute pain levels
100mm Visual Analogue Scale (VAS) with the end-points "no pain" and "worst pain possible" | Study Visit 4 (Week 12)
  * It is a reliable and valid measure of self-reported pain intensity
  * VAS is administered before and after intervention to evaluate acute pain levels

OTHER OUTCOMES:
Patient reported Verbal Compliance Ratings | Study Visit 2 (Week 4)
  Patient reported Verbal Compliance Ratings towards the use of the foot orthosis fitted and other standard podiatry management using a verbal compliance ratings form administered by the investigators during the study visit will be carried out.
Patient reported Verbal Compliance Ratings | Study Visit 3 (Week 8)
  Patient reported Verbal Compliance Ratings towards the use of the foot orthosis fitted and other standard podiatry management using a verbal compliance ratings form administered by the investigators during the study visit will be carried out.
Patient reported Verbal Compliance Ratings | Study Visit 4 (Week 12)
  Patient reported Verbal Compliance Ratings towards the use of the foot orthosis fitted and other standard podiatry management using a verbal compliance ratings form administered by the investigators during the study visit will be carried out.
Patient Satisfaction Ratings | Study Visit 2 (Week 4)
  Collection of Patient Satisfaction Ratings using a verbal compliance ratings form administered by the investigators during the study visit will be carried out.
Patient Satisfaction Ratings | Study Visit 3 (Week 8)
  Collection of Patient Satisfaction Ratings using a verbal compliance ratings form administered by the investigators during the study visit will be carried out.
Patient Satisfaction Ratings | Study Visit 4 (Week 12)
  Collection of Patient Satisfaction Ratings using a verbal compliance ratings form administered by the investigators during the study visit will be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Guan Ng, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Foot Care and Limb Design Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manoli A 2nd, Graham B. The subtle cavus foot, "the underpronator". Foot Ankle Int. 2005 Mar;26(3):256-63. doi: 10.1177/107110070502600313. PMID 15766431
- [Background] Chilvers M, Manoli A 2nd. The subtle cavus foot and association with ankle instability and lateral foot overload. Foot Ankle Clin. 2008 Jun;13(2):315-24, vii. doi: 10.1016/j.fcl.2008.01.003. PMID 18457776
- [Background] Desai SN, Grierson R, Manoli II A. The cavus foot in athletes: fundamentals of examination and treatment. Operative Techniques in Sports Medicine. 2010 Mar 1;18(1):27-33.
- [Background] Beals TC, Manoli A. The'peek-a-boo'heel sign in the evaluation of hindfoot varus. The Foot. 1996;4(6):205-6.
- [Background] Coleman SS, Chesnut WJ. A simple test for hindfoot flexibility in the cavovarus foot. Clin Orthop Relat Res. 1977 Mar-Apr;(123):60-2. No abstract available. PMID 852192
- [Background] Burns J, Crosbie J, Ouvrier R, Hunt A. Effective orthotic therapy for the painful cavus foot: a randomized controlled trial. J Am Podiatr Med Assoc. 2006 May-Jun;96(3):205-11. doi: 10.7547/0960205. PMID 16707631
- [Background] Burns J, Landorf KB, Ryan MM, Crosbie J, Ouvrier RA. Interventions for the prevention and treatment of pes cavus. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD006154. doi: 10.1002/14651858.CD006154.pub2. PMID 17943889
- [Background] LoPiccolo M, Chilvers M, Graham B, Manoli A 2nd. Effectiveness of the cavus foot orthosis. J Surg Orthop Adv. 2010 Fall;19(3):166-9. PMID 21086930
- [Background] Abbasian A, Pomeroy G. The idiopathic cavus foot-not so subtle after all. Foot Ankle Clin. 2013 Dec;18(4):629-42. doi: 10.1016/j.fcl.2013.08.004. PMID 24215829
- [Background] Landorf KB, Twyford GN, Cotchett MP, Whittaker GA. Revised minimal important difference values for the visual analogue scale and Foot Health Status Questionnaire when used for plantar heel pain. J Foot Ankle Res. 2024 Dec;17(4):e70021. doi: 10.1002/jfa2.70021. PMID 39682003